CLINICAL TRIAL: NCT03581500
Title: Hyperpolarized 13-C-Pyruvate Magnetic Resonance Spectroscopic Imaging Reproducibilty Pilot in Patients With Prostate Cancer
Brief Title: Hyperpolarized Carbon C 13 Pyruvate Magnetic Resonance Spectroscopic Imaging in Predicting Treatment Response in Patients With Prostate Cancer
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Committee could not find that the regulatory approval are met to re-approve this study.
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2017-0403; NCI-2018-01096 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2017-0403 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2018-06-27; First posted 2018-07-10 (Actual); Last update posted 2025-04-23 (Actual); Status verified 2024-10

CONDITIONS: Prostate Adenocarcinoma; PSA Level Greater Than Ten; Stage IIB Prostate Cancer AJCC v8; Stage III Prostate Cancer AJCC v8; Stage IIIA Prostate Cancer AJCC v8; Stage IIIB Prostate Cancer AJCC v8; Stage IIIC Prostate Cancer AJCC v8; Stage IV Prostate Cancer AJCC v8; Stage IVA Prostate Cancer AJCC v8; Stage IVB Prostate Cancer AJCC v8
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Diagnostic (hyperpolarized carbon C 13 pyruvate MRSI) (Experimental): Patients receive hyperpolarized carbon C 13 pyruvate IV over 10-20 seconds and undergo MRSI over 2-3 minutes at 6 and 8 weeks.
  Interventions: Drug: Hyperpolarized Carbon C 13 Pyruvate; Procedure: Magnetic Resonance Spectroscopic Imaging

INTERVENTIONS:
Drug: Hyperpolarized Carbon C 13 Pyruvate — Given IV
  Other Names: Hyperpolarized 13C-Pyruvate; Hyperpolarized Pyruvate (13C)
Procedure: Magnetic Resonance Spectroscopic Imaging — Undergo MRSI
  Other Names: 1H- Nuclear Magnetic Resonance Spectroscopic Imaging; 1H-nuclear magnetic resonance spectroscopic imaging; Magnetic Resonance Spectroscopy; MRS; MRS Imaging; MRSI; Proton Magnetic Resonance Spectroscopic Imaging

SUMMARY:
This phase II trial studies how well hyperpolarized carbon C 13 pyruvate magnetic resonance spectroscopic imaging works in predicting treatment response in patients with prostate cancer. Hyperpolarized carbon C 13 pyruvate magnetic resonance spectroscopic imaging may help to accurately predict how prostate cancer patients will respond to standard therapy (abiraterone and apalutamide).

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To assess reproducibility of quantitative spectroscopic and imaging parameters in hyperpolarized 13-C pyruvate magnetic resonance spectroscopic imaging (MRSI), including key performance indicator (kpl), which assesses the rate of conversion of 13-C pyruvate to 13-C lactate in the tissue of interest, using a test-retest study design.

SECONDARY OBJECTIVE:

I. To provide initial assessment of the sensitivity and specificity of hyperpolarized 13-C-pyruvate MRSI performed pre-therapy for detecting high risk localized prostate cancer.

OUTLINE:

Patients receive hyperpolarized carbon C 13 pyruvate intravenously (IV) over 10-20 seconds and undergo MRSI over 2-3 minutes at 6 and 8 weeks.

After completion of study, patients are followed up at 1 day and then for up to 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Biopsy proven high risk prostate adenocarcinoma, or de novo metastatic previously untreated naive prostate cancer (patients who have initiated gonadotrophin releasing hormone [Lhrh] analog or antagonist within the past 4 weeks are eligible)
* Gleason >= 8 OR Gleason 7 + >= cT2b + prostate specific antigen (PSA) > 10 ng/ml
* Prior prostate biopsy must have been performed at least 4 weeks prior

Exclusion Criteria:

* Contraindication to MRI
* Estimated glomerular filtration rate (eGFR) < 30
* Allergy to gadavist intravenous contrast
* History of cardiac arrhythmia
* Since they do not get prostate cancer, women are excluded; thus, pregnancy is not an issue

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-02-06 (Actual); Primary Completion 2024-10-16 (Actual); Study Completion 2024-10-16 (Actual)

PRIMARY OUTCOMES:
Reproducibility of the key performance indicator | Up to 3 years

SECONDARY OUTCOMES:
Sensitivity assessed by comparison to biopsy | Up to 3 years
  The location of signal by hyperpolarized 13-C-pyruvate will be compared to location of tumor at biopsy or if available, follow-up surgical pathology in patients who did not receive interval additional prostate directed therapy, such as hormonal or radiation therapy.
Specificity assessed by comparison to biopsy | Up to 3 years
  The location of signal by hyperpolarized 13-C-pyruvate will be compared to location of tumor at biopsy or if available, follow-up surgical pathology in patients who did not receive interval additional prostate directed therapy, such as hormonal or radiation therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Tharakeswara Bathala, MBBS,MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org